CLINICAL TRIAL: NCT03281018
Title: Exploratory Study of the Impact of a Preoperative Formal Hypnosis Session on Perioperative Anxiety Among Female Patients Hospitalised for Hysterectomy Due to Pelvic Gynecological Cancer
Brief Title: Preoperative Hypnosis in Gynecology
Acronym: HYPPOGYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2016/18
Record Dates: First submitted 2017-09-01; First posted 2017-09-13 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Gynecological Cancer
Keywords: hypnosis; preoperative anxiety; hysterectomy; hospitalisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): Caregiver Accompaniment Time (CAT) + preoperative hypnosis session (experimental arm): The hypnosis session is performed by a nurse trained in medical hypnosis; this interview lasts approximately one hour and is carried out 5 to 15 days before the hospitalisation. During the hypnosis session, the patient is free to choose what issues she wants to address. The patient will then go from a state of ordinary consciousness to a modified state of consciousness. This state will allow her to activate her own resources to handle difficulties, especially anxiety. Using a post-hypnotic suggestion, the patient will be able to revisit her work at any time she needs
  Interventions: Behavioral: Caregiver Accompaniment Time (CAT) + preoperative hypnosis session
- Control (CAT) (No Intervention): CAT is performed in routine care for all patients after the announcement of the illness by a trained nurse, if possible on the same day as the consultation or before the consultation of anesthesia. This is an interview of approximately 45 minutes to listen to the patient, to answer her questions and to re-explain the information delivered to her. The patient will tackle the history of the disease and then the treatment, this time dedicated evolves according to the desire of the patient and her ability to accept the disease. The patient can express her feelings, then the family circle is evoked talking about the resource persons and the future. The purpose of this interview is to obtain the autonomy of the patient by the setting up of supportive care

INTERVENTIONS:
Behavioral: Caregiver Accompaniment Time (CAT) + preoperative hypnosis session — The hypnosis session is performed by a nurse trained in medical hypnosis; this interview lasts approximately one hour and is carried out 5 to 15 days before the hospitalisation. During the hypnosis session, the patient is free to choose what issues she wants to address. The patient will then go from a state of ordinary consciousness to a modified state of consciousness. This state will allow her to activate her own resources to handle difficulties, especially anxiety. Using a post-hypnotic suggestion, the patient will be able to revisit her work at any time she needs
  Arms: Interventional arm

SUMMARY:
The research hypotheses that preoperative formal hypnosis session reduces perioperative anxiety among women undergoing a hysterectomy for pelvic gynecological cancer. The key objective is to estimate the effect of preoperative hypnosis on preoperative anxiety among this population

DETAILED DESCRIPTION:
Anxiety is present preoperatively in 40% of patients. The operated subjects are on average 20% more anxious than the general population, according to a study of 2013. Cancer as well as surgery modifying the body pattern and impairing femininity are risk factors for preoperative anxiety. Recent work in both children and adults has shown that significant levels of preoperative anxiety increase the risk of postoperative complications and the occurrence of postoperative emotional and behavioral disorders. The consequences of hysterectomy increase patients' anxiety, for fear of affecting femininity, and the modification of the body regimen. The prevention of preoperative anxiety in such population is therefore a major issue.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18yrs with pelvic gynecological cancer (endometrium, cervix, ovary),
* at any stage of the disease;
* patient coming for anesthesia consultation before hysterectomy,
* informed signed consent,
* patient affiliated to or beneficiary of social security.

Exclusion Criteria:

* patient <18yrs,
* patient with a pelvic gynecological cancer that does not require hysterectomy;
* patient with psychiatric history or a depressive syndrome;
* deaf patient (deafness makes the hypnosis session impossible),
* patient under legal protection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
evolution of anxiety | 1 month after the surgery
  visual analog scale (from 0, no anxiety to 10, extreme anxiety)

SECONDARY OUTCOMES:
pain | The day of the consultation with anesthesist, the day before the surgery, 2 days, an average of 12 days, and 1 month after the surgery
  numerical scale of pain (from 0, no pain, to 10, extreme pain)
nausea and vomiting | 2 days, an average of 12 days, and 1 month after the surgery
  frequency and intensity through an interview with a nurse
concomitant medication | The day of the consultation with anesthesist, the day before the surgery, 2 days, an average of 12 days, and 1 month after the surgery
  concomitant medication within anxiolytic, antalgic, and/or antiemetic pharmaceutical classes (yes/no)
medical history | The day of the consultation with anesthesist
  chronic pathologies (e.g. arterial hypertension, type 2 diabetes) (yes/no)
length of hospital stay | an average of 12 days after the surgery
hypnosis intervention feasibility (composite outcome) | after the hypnosis session (average of 1 week before the surgery)
  Compliance with the formal Hypnosis session checklist (Installation, pre-session interview, kinesthetic induction, dissociation, deepening, post-hypnotic suggestions and anchoring, return to normal wakefulness)
  Other factors: proportion of refusals, proportion of abandoned, proportion of lost sight

CONTACTS AND LOCATIONS:
Overall Officials: Jennie SOURZAC, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU Bordeaux, Bordeau, France